CLINICAL TRIAL: NCT00528268
Title: Prospective Phase I/II Study to Evaluate Effects of Sodium Phenylbutyrate in Pre-symptomatic Infants With Spinal Muscular Atrophy
Brief Title: Study to Evaluate Sodium Phenylbutyrate in Pre-symptomatic Infants With Spinal Muscular Atrophy
Acronym: STOPSMA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22183; 1R01HD054599-01 (NIH)
Record Dates: First submitted 2007-09-10; First posted 2007-09-12 (Estimated); Results first posted 2015-07-03 (Estimated); Last update posted 2025-02-28 (Actual); Status verified 2017-06

CONDITIONS: Spinal Muscular Atrophy
Keywords: Spinal Muscular Atrophy; SMA; Sodium Phenylbutyrate
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — 4-phenylbutyric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cohort 1 (Active Comparator): Treatment with sodium phenylbutyrate; age < 3 months; history of sibling(s) with type I SMA; SMN2 dosage < 3 copies
  Interventions: Drug: Sodium phenylbutyrate
- cohort 2 (Active Comparator): Treatment with sodium phenylbutyrate; age < 6 months; history of sibling(s) with type II SMA; SMN2 dosage < 4 copies
  Interventions: Drug: Sodium phenylbutyrate

INTERVENTIONS:
Drug: Sodium phenylbutyrate — Sodium phenylbutyrate is dispensed as a powder, 450-600 mg/kg/day, divided into four doses. For cohort 1, treatment and monitoring continues for 18 months. For cohort 2, treatment and monitoring continues for 24 months.
  Other Names: NaPB

SUMMARY:
In this single-center trial, we will evaluate the effects of NaPB on presymptomatic Spinal Muscular Atrophy (SMA) type I (cohort 1)and presymptomatic SMA type II (cohort 2) infants. A variety of outcome measures will be performed at each study visit to follow the course of the disease. Total duration of the study for type I infants will be 18 months, for type II infants, 24 months.

DETAILED DESCRIPTION:
Perform a phase I/II study to evaluate effects of sodium phenylbutyrate (NaPB) in a cohort of presymptomatic infants, predicted to develop either SMA type 1 or SMA type 2 given genotype and family history of an older sibling with the respective SMA type. Primary outcomes: 1) to collect additional safety and pharmacokinetic data in neonates and young infants administered NaPB within the dosing guidelines already in use for urea cycle disorder therapy, and 2) to determine possible benefit of early treatment intervention with regard to status of denervation and functional motor status at specific time points for which we have matched natural history data to perform a comparison between cohorts and between each cohort and participants from our natural history database matched for age, SMN2 dosage and gender.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory documentation of homozygous absence of SMN1 exon 7.
* Confirmation of no more than 3 SMN2 copies for cohort 1; no more than 4 copies for cohort 2.
* Family history of affected sibling with SMA type I for cohort 1 and SMA type II for cohort 2.
* Age ≤ 3 months, cohort 1; Age ≤ 6 months, cohort 2.
* Written informed consent of parents/guardian.
* Laboratory results demonstrating normal values for age.

Exclusion Criteria:

-Evidence of hepatic insufficiency, renal insufficiency, edema with sodium retention, known seizure disorder, urea cycle disorder, cardiac arrhythmia, congenital heart defect, hypertension, significant central nervous system (CNS) impairment, or neurodegenerative or neuromuscular disease other than SMA.

History of allergy/sensitivity to sodium phenylbutyrate (NaPB).

* Use of NaPB within 30 days of study entry.
* Serious illness requiring hospitalization ≤ 14 days prior to study entry.
* Use of medications intended for the treatment of SMA including riluzole, valproic acid, hydroxyurea, oral use of albuterol, NaPB, butyrate derivatives, creatine, growth hormone, anabolic steroids, probenecid, oral or parenteral use of corticosteroids at entry, or agents anticipated to increase or decrease muscle strength or agents with presumed histone deacetylase (HDAC) inhibition within 30 days prior to study entry.
* Unwillingness to travel for study assessments.

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2007-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Swoboda, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon request, to include the following outcomes data: 1) degree of denervation as measured over time by maximum ulnar compound muscle action potential amplitude (both cohorts); % of patients who die or require > 16 hours ventilator support for more than 4 weeks by 18 months of age (cohort I); % of patients who achieve independent sitting for at least 30 seconds (cohort I); % of patient who achieve independent ambulation by 2 years of age (cohort II)

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Family history of SMA type I 0-3 months old Confirmation of no more than 3 SMN2 copies
  Sodium phenylbutyrate (NaPB): The powder form of the drug will be dispensed. The target NaPB dosing is 450-600 mg/kg/day, divided into four doses. For cohort 1, we propose to continue treatment for 18 months. For cohort 2, we propose to continue treatment for 24 months.
- Cohort 2: Family history of SMA type II 0-6 months old Confirmation of no more than 4 SMN2 copies
  Sodium phenylbutyrate (NaPB): The powder form of the drug will be dispensed. The target NaPB dosing is 450-600 mg/kg/day, divided into four doses. For cohort 1, we propose to continue treatment for 18 months. For cohort 2, we propose to continue treatment for 24 months.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 6 | 8
Completed | 5 | 7
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 8 | 14
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Sodium Phenylbutyrate in Neonates and Infants With SMA
Description: The number of participants able to achieve specific developmental milestones, such as sitting unsupported or walking independently, during the study period.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 6 | 8
Participants
  Able to sit unsupported | 1 | 8
  Able to walk independently | 0 | 1

ADVERSE EVENTS:
Arm/Group | Cohort 1 | Cohort 2
Serious Adverse Events (participants affected / at risk) | 6/6 | 7/8
Other Adverse Events (participants affected / at risk) | 6/6 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=6) | Cohort 2 (N=8)
Daily Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
GE Reflux (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 3 (4) | 0 (0)
Anemia of Chronic Disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lung Collapse (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
G-tube (Gastrointestinal disorders) | 3 (3) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Failure to swallow (Gastrointestinal disorders) | 1 (1) | 0 (0)
ALTE (General disorders) | 1 (1) | 0 (0)
Nystagmus (Nervous system disorders) | 1 (1) | 0 (0)
Dehydration (General disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Recurrent Reflux (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 4 (8) | 1 (2)
Increased Secretions (General disorders) | 1 (1) | 1 (1)
Death (General disorders) | 1 (1) | 1 (1)
Medication Error (Investigations) | 0 (0) | 1 (1)
Lethargy (General disorders) | 0 (0) | 2 (2)
Foot and Mouth Disese (Infections and infestations) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=6) | Cohort 2 (N=8)
Serous Otitis Media Bilateral (Infections and infestations) | 4 (6) | 3 (4)
Eye Infection (Infections and infestations) | 1 (1) | 1 (2)
Upper Respiratory Infection (Infections and infestations) | 2 (2) | 3 (4)
Flu symptoms (Infections and infestations) | 2 (2) | 5 (10)
Rhinitis (Infections and infestations) | 2 (2) | 1 (1)
Encephalopathy (Infections and infestations) | 1 (1) | 0 (0)
Swelling (General disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Thrush (Infections and infestations) | 1 (1) | 0 (0)
Left Wrist drop (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Increased Secretion (General disorders) | 1 (1) | 0 (0)
Gasteroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Increased Heart Rate (Investigations) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Spontaneous Drop in Saturations (Investigations) | 1 (1) | 0 (0)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Zinc Deficiency (Investigations) | 1 (1) | 0 (0)
Reflux (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hand foot mouth disease (Infections and infestations) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
strep throat (Infections and infestations) | 0 (0) | 1 (1)
Unable to Eat (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infected Cyst (Infections and infestations) | 0 (0) | 1 (1)
Placement of bilateral ear tubes (Ear and labyrinth disorders) | 0 (0) | 1 (1)
H1N1 (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Sinus Infection (Infections and infestations) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Blank Stare (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes